CLINICAL TRIAL: NCT00359450
Title: A Three Cohort Phase II Trial of BMS-275183 Given Orally on a Twice Weekly Schedule in Pretreated Locally Advanced or Metastatic NSCLC Patients
Brief Title: Study of BMS-275183 in Patients With Pretreated Locally Advanced or Metastatic NSCLC (Non Small Cell Lung Cancer)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA165-026; EUDRACT: 2005-005099-33
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2007-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Locally advanced or metastatic non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — BMS-275183; taxane

INTERVENTIONS:
Drug: BMS-275183 (oral taxane)

SUMMARY:
BMS-275183 given orally twice weekly to patients pretreated for locally advanced or metastatic NSCLC will show anti-tumor activity in any of the 3 separate cohorts of the patients enrolled:

* Cohort I: Patients previously treated with one taxane containing regimen.
* Cohort II: Patients previously treated with a platinum based but non-taxane containing regimen.
* Cohort III: Patients previously treated with both a chemotherapy regimen and one EGFR-TKI (epidermal growth factor receptor-tyrosine kinase inhibitor) compound.

Patients in cohorts I and II should have not been treated with a prior EGFR-TKI compound. Prior treatment with a VEGFR (vascular endothelial growth factor receptor) inhibitor compound is allowed for all the patients provided that the VEGFR inhibitor is not also an EGFR inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age >= 18 years
* Subjects with histologically or cytologically confirmed locally advanced or metastatic NSCLC who failed only one prior chemotherapy regimen.

Exclusion Criteria:

* Concomitant medication with a cytochrome P450 (CYP) 3A4 inhibitor or inducer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186
Dates: Start 2006-07; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To assess efficacy of BMS-275183 in pretreated NSCLC patients as measured by the tumor response rate

SECONDARY OUTCOMES:
To further characterize the qualitative and quantitative toxicities of BMS-275183 in the same patient population
Assess the response duration
Assess the progression free survival time
Assess the overall survival time
Assess the pharmacokinetics (PK) of BMS-275183

CONTACTS AND LOCATIONS:
Locations (30):
- United States (4):
  - Local Institution, Burlington, Massachusetts
  - Local Institution, St Louis, Missouri
  - Local Institution, Morganton, North Carolina
  - Local Institution, Cleveland, Ohio
- Belgium (2):
  - Local Institution, Charleroi
  - Local Institution, Leuven
- Canada (4):
  - Local Institution, Montreal, Ontario
  - Local Institution, Thunder Bay, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Saint-Jérôme, Quebec
- France (6):
  - Local Institution, Belfort
  - Local Institution, Besançon
  - Local Institution, Poitiers
  - Local Institution, Saint-Herblain
  - Local Institution, Strasbourg
  - Local Institution, Tours
- Italy (4):
  - Local Institution, Napoli
  - Local Institution, Orbassano Torino
  - Local Institution, Perugia
  - Local Institution, Roma
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Maastricht
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Madrid
- United Kingdom (6):
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, Glasgow, Central
  - Local Institution, Plymouth, Devon
  - Local Institution, London, Greater London
  - Local Institution, Northwood, Middlesex
  - Local Institution, Oxford, Oxfordshire